CLINICAL TRIAL: NCT01187004
Title: Extracardiac Complications After Cardiopulmonary by Pass in Cardiac Surgery
Brief Title: Extracardiac Complications After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Daniela Pasero, MD, University of Turin, Italy
Other Study IDs: 82755
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Results first posted 2012-01-06 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Acute Lung Injury; Sepsis; Infections; Acute Kidney Injury
MeSH Terms: conditions — Acute Lung Injury; Sepsis; Infections; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute Lung Injury (ALI): patients who might develop acute lung injury (ALI) after cardiac surgery with cardiopulmonary by pass

SUMMARY:
Hypothesis of the study is that patients undergoing major cardiac surgery can develop extracardiac complications correlated to cardiopulmonary by pass.

DETAILED DESCRIPTION:
To find out which are the main peri operative predictors of acute lung injury and other extracardiac complications, such as kidney injury, that prolonged Intensive Care Unit (ICU) length of stay after cardiac surgery. The main goal is to evaluate whether mechanical ventilation, in particular tidal volume, can be predictor of acute lung injure in this kind of patients.

ELIGIBILITY:
Inclusion Criteria:

* cardiac intervention with cardiopulmonary by pass, age > 18 years old

Exclusion Criteria:

* off-pump surgery, heart and lung transplantations, patients on mechanical ventilation before intervention or admitted to Intensive Care Unit (ICU) before intervention.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing major cardiac surgery with cardiopulmonary by pass
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Rinaldi, MD, Study Chair — San Giovanni Battista Hospital, University of Turin
Locations (1):
- Cardiac Intensive Care Unit, San Giovanni Battista Hospital, Turin, Italy, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled all patients undergoing a cardiac surgery intervention on cardiopulmonary by pass (CPB)
Pre-assignment Details: Patients were excluded for: Intensive Care Unit - Length of stay (ICU-LOS)<24h, age < 18 yrs old; mechanical ventilation before surgery; Acute Lung Injury (ALI) at the admission to Intensive Care Unit (ICU); heart and lung transplant
Groups:
- Acute Lung Injury (ALI) Group: patients who develop acute lung injury (ALI) after cardiac surgery with cardiopulmonary by pass
- Control Group: patients who don't develop acute lung injury after cardiac surgery with cardiopulmonary by pass
Period: Overall Study
Arm/Group | Acute Lung Injury (ALI) Group | Control Group
Started | 20 | 144
Completed | 20 | 144
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Lung Injury (ALI) Group | Control Group | Total
Number analyzed (Participants) | 20 | 144 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 57 | 64
  >=65 years | 13 | 87 | 100
Age Continuous [Mean (Standard Deviation); unit: years] | 69 (10) | 65 (14) | 66 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 38 | 47
  Male | 11 | 106 | 117
Region of Enrollment [Number; unit: participants]
  Italy | 20 | 144 | 164

OUTCOME MEASURES:

1. Primary Outcome: Acute Lung Injury After Cardiac Surgery
Description: to evaluate the incidence of acute lung injury (ALI) in patients undergoing cardiac surgery with cardiopulmonary by pass and to identify the main predictors.Diagnosis of Acute Lung Injury (ALI) was made according to the American-European Consensus conference criteria, including acute onset, PaO2 /FiO2 <300 regardless of Positive End Expiratory Pressure (PEEP) level, bilateral and diffuse opacities on chest radiograph, absence of left ventricular failure, or history of lung disease.
Time Frame: at seven days after intervention
Population: Patients consecutively admitted to the cardiac Intensive Care Unit (cICU) after cardiac surgery on cardiopulmonary by pass (CPB), during a time frame of two years.The analysis was per protocol, to identify the predictors of acute lung injury after cardiac surgery.
Measure: Number; unit: participants
Groups:
- Acute Lung Injury: Patients who developed acute lung injury (ALI) after cardiac surgery and during mechanical ventilation
Arm/Group | Acute Lung Injury
Number analyzed (Participants) | 164
participants | 20 [6 to 16]
Statistical Analysis 1: Comparison: Acute Lung Injury; Our hypothesis was that mechanical ventilation with large tidal volume might represent a risk factor for acute lung injury in patients undergoing cardiopulmonary bypass; Test type: Superiority or Other; p < 0.05, Regression, Logistic; significant level for inclusion at the univariate analysis was p<0.05; Odds Ratio (OR) = 1

2. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay
Description: If extracardiac complications, especially acute lung injury, prolonged Intensive Care Unit (ICU) length of stay due to longer mechanical ventilation.
Time Frame: at 28 days
Population: The analysis of the Intensive Care Unit (ICU) length of stay was done on all the patients included in the study. We want to evaluate if the development of acute lung injury prolongs the intensive care unit length of stay.ICU length of stay was calculated up to 28 days,and patients who died before were considered as having the maximum value
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- ICU-LOS in Patients Developing ALI: Intensive care unit length of stay in patients developing acute lung injury. ICU length of stay was calculated up to 28 days, and patients who died before were considered as having the maximum value
- Control Group: patients who didn't develope ALI. ICU length of stay was calculated up to 28 days, and patients who died before were considered as having the maximum value
Arm/Group | ICU-LOS in Patients Developing ALI | Control Group
Number analyzed (Participants) | 20 | 144
days | 22 (54) [4 to 26] | 2 [1 to 26]
Statistical Analysis 1: Comparison: ICU-LOS in Patients Developing ALI vs Control Group; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.199, 95% CI 2-sided [1.129 to 1.272]

ADVERSE EVENTS:
Arm/Group | Acute Lung Injury (ALI) Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/144
Other Adverse Events (participants affected / at risk) | 0/20 | 0/144

LIMITATIONS AND CAVEATS:
The main limitation of the trial was the observational nature and the relatively small number of patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No